CLINICAL TRIAL: NCT04081831
Title: Effectiveness of Low-dose Aspirin in Gastrointestinal Cancer Prevention - Hong Kong
Brief Title: Effectiveness of Low Dose Aspirin in Decreasing the Chance Getting Stomach and Intestine Cancer
Acronym: ENgAGE-HK
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20319
Record Dates: First submitted 2019-07-30; First posted 2019-09-09 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Gastrointestinal Cancer
Keywords: Esophageal cancer; Gastric cancer; Colorectal cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New-users of Low-dose aspirin (exposed group): New-users of low-dose aspirin is defined as patients who did not receive any prescriptions of low-dose aspirin one year prior to the index date.
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- Users of Paracetamol (non-exposed group): Users of Paracetamol is defined as patients who receive first prescription of paracetamol during the study period. Since the patients receiving low-dose aspirin are potentially less healthy compared to non-users of aspirin, patients receiving paracetamol as the control group can minimise healthy user bias.

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin, BAYE4465) — Follow clinical administration
  Groups: New-users of Low-dose aspirin (exposed group)

SUMMARY:
In this study, researchers wanted to learn more about the effect of Aspirin taken as low dose (75 - 300 mg) in preventing stomach, colorectal and esophagus cancer. The researchers were interested in the effect by duration of aspirin use and the effect on the time since aspirin intake has been stopped in preventing stomach, colorectal and esophagus cancer. In addition, the study also looked into the time patients survived after being diagnosed (survival rate) with cancer and number of cancer patients who died (case fatality rate). The study was based on an electronic database managed by the Health Authority in Hong Kong containing anonymized clinical information of patients living in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

- Received prescription of either low-dose aspirin (75-300 mg) or paracetamol monotherapy during enrolment period.

Exclusion Criteria:

* Received prescription of aspirin monotherapy or combination one year prior to the index date
* Recorded diagnoses of any type of cancer before the index date
* Recorded procedures of colectomy, gastrectomy prior to the index date
* Age < 40 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 40 years who received low dose aspirin (75-300 mg) or paracetamol between 1st January 2004 and 31st December 2008 will be identified from CDARS (Clinical Data Analysis and Reporting System). CDARS is an electronic clinical database which is managed by the Hospital Authority (HA). More than seven million Hong Kong citizens have access to public healthcare services provided by HA.
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Incidence rate ratio of colorectal cancer among users of low-dose-aspirin (exposed) and users of paracetamol monotherapy (non-exposed) | Retrospective analysis between 1st January 2004 and 31st December 2008
  Ratio of incidence (per 10,000 person years) among users of low-dose-aspirin (exposed) and users of paracetamol monotherapy (non-exposed)
Incidence rate ratio of gastric cancer among users of low-dose-aspirin (exposed) and users of paracetamol monotherapy (non-exposed) | Retrospective analysis between 1st January 2004 and 31st December 2008
  Ratio of incidence (per 10,000 person years) among users of low-dose-aspirin (exposed) and users of paracetamol monotherapy (non-exposed)
Incidence rate ratio of esophageal cancer among users of low-dose-aspirin (exposed) and users of paracetamol monotherapy (non-exposed) | Retrospective analysis between 1st January 2004 and 31st December 2008
  Ratio of incidence (per 10,000 person years) among users of low-dose-aspirin (exposed) and users of paracetamol monotherapy (non-exposed)

SECONDARY OUTCOMES:
Duration of aspirin use | Retrospective analysis between 1st January 2004 and 31st December 2008
  Minimum duration of aspirin use to confer the protective effects in preventing colorectal, gastric and esophageal cancer
Risk of colorectal, gastric and esophageal cancer after discontinuation of aspirin use | Retrospective analysis between 1st January 2004 and 31st December 2008
  Logistic regression will be conducted based on nested case-control study with stratification on the recency of exposure with current use, past use, and distant use of aspirin.
Case-fatality and survival rate | Retrospective analysis between 1st January 2004 and 31st December 2008
  For colorectal cancer, gastric or oesophageal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.